CLINICAL TRIAL: NCT04337710
Title: Exclusive Enteral Nutrition in Preterm Neonates- A Randomized Controlled Trial
Brief Title: Exclusive Enteral Nutrition in Preterm Neonates
Acronym: ENACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300004922
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Premature; Infant, Light-for-dates; Enteral Feeding Intolerance
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive Enteral Nutrition (Experimental): This group will receive enteral feeding volumes at a rate of 60-80 ml/kg/day starting within the first 24 hours after birth. Volumes will increase by 20-30 ml/kg/day until intake is 150ml/kg/day.
  Interventions: Procedure: Exclusive Enteral Nutrition
- Progressive Enteral Nutrition (Active Comparator): This group will receive enteral feeding volumes at a rate of 20-30 ml/kg/day starting within the first 24 hours after birth. Volumes will increase by 20-30 ml/kg/day until intake is 150ml/kg/day.
  Interventions: Procedure: Progressive Enteral Nutrition

INTERVENTIONS:
Procedure: Exclusive Enteral Nutrition — Mom's milk or donor milk at 60-80 ml/kg/day after randomization within the first 24 hours.
  Arms: Exclusive Enteral Nutrition
Procedure: Progressive Enteral Nutrition — Mom's milk or donor milk at 20-30 ml/kg/day after randomization within the first 24 hours.
  Arms: Progressive Enteral Nutrition

SUMMARY:
To test the hypothesis that early exclusive enteral nutrition with the minimal use of parenteral nutrition will improve preterm infants' nutritional outcomes when compared to delayed progression of enteral nutrition and prolonged use of parenteral nutrition.

DETAILED DESCRIPTION:
Qualifying participants will be randomly assigned to one of two study groups: 1) Exclusive Enteral Feeds or 2) Progressive Enteral Feeds with supplemental parenteral nutrition. Regardless of study group assignment, donor human milk will be offered if the mother's expressed breast milk is not enough to complete the intervention as assigned.

Intervention group: Feeds will be initiated with a target volume of 60-80 ml/kg/day and then advanced by 20-30 ml/kg/day until the total volume of 150ml/kg/day is achieved.

Control group: Enteral feeds will be initiated with a target volume of 20-30 ml/kg/day and then advanced by 20-30 ml/kg/day until the total volume of 150 ml/kg/day is achieved.

If parent agrees, stool "dirty" diapers will be collected 2 times during this study.

One time around the time of birth and one time at 28 days or discharge (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 and 32 weeks of gestation

Exclusion Criteria:

* Intrauterine growth restriction (birth weight < 10th percentile)
* Major congenital or chromosomal anomalies
* Terminal illness in which decisions to withhold or limit support have been made

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of days of full enteral feeding (150ml/kg/day) in the first 28 days after birth | Birth to 28 days
  Days of full feeds in the first 28 days after birth

SECONDARY OUTCOMES:
Time to establish full enteral feeding | Birth to 28 days
  Time interval between birth and full enteral feeding at 150ml/kg/day
Number of episodes of feeding intolerance | Birth to 28 days
  Interruption or cessation of enteral feeds for a period greater than 12 hours for abnormal abdominal examination
Number of days receiving parenteral nutrition and IV fluids | Birth to 28 days
Number of days receiving central line access | Birth to 28 days
Number of episodes of culture proven sepsis | Birth to 60 days or discharge, whichever occurs first
  Positive blood cultures
Number of participants with diagnosis of necrotizing enterocolitis | Birth to 60 days or discharge, whichever occurs first
  Diagnosis of necrotizing enterocolitis stage 2 or 3
Number of participants with diagnosis of intestinal perforation | Birth to 14 days
  Pneumoperitoneum on abdominal radiograph
Death | Birth to 60 days
Weight | Birth to 60 days
  Weekly measurements of weight in g
Length | Birth to 60 days
  Weekly measurements of length in cm
Head circumference | Birth to 60 days
  Weekly measurements of head circumference in cm
Duration of hospital stay in days | Birth to 60 days

OTHER OUTCOMES:
Intestinal microbiome profile | At postnatal day 14
  Determined by molecular analyses of bacterial fragments in fecal samples
Fat-free mass z score | At postnatal day 14
  Determined by air-displacement plethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Shukla, MD, Study Chair — University of Alabama at Birmingham; Ariel Salas, MD, MSPH, Study Director — University of Alabama at Birmingham; Jacqueline Razzaghy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Razzaghy J, Shukla VV, Gunawan E, Reeves A, Nguyen K, Salas AA. Early and exclusive enteral nutrition in infants born very preterm. Arch Dis Child Fetal Neonatal Ed. 2024 Jun 19;109(4):378-383. doi: 10.1136/archdischild-2023-325969. PMID 38135494
- [Derived] Salas AA, Stewart CJ, Young GR. Early gut microbiome composition of very preterm infants randomised to receive human milk volumes of 60 ml/kg/day or more within the first 36 hours after birth. Pediatr Res. 2025 Oct 2. doi: 10.1038/s41390-025-04456-5. Online ahead of print. PMID 41034647
- See also: Commentary — https://neonatalnutritionresearch.com/f/our-journey-investigating-early-exclusive-enteral-nutrition